CLINICAL TRIAL: NCT00760175
Title: A Randomized, Controlled Trial Comparing Intradermal Versus Intramuscular Trivalent Influenza Vaccine in Adult Lung Transplant Recipients
Brief Title: Intradermal Versus Intramuscular Trivalent Influenza Vaccine in Adult Lung Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: University of Lausanne Hospitals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 7407
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Influenza Virus; Influenza Vaccine
Keywords: Lung transplant Recipients; Vaxigrip
MeSH Terms: conditions — Influenza, Human | interventions — vaxigrip; Influenza Vaccines

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intradermal (Active Comparator)
  Interventions: Biological: Vaxigrip (Aventis-Pasteur Canada)
- intramuscular (Active Comparator)
  Interventions: Biological: Vaxigrip (Aventis-Pasteur Canada)

INTERVENTIONS:
Biological: Vaxigrip (Aventis-Pasteur Canada) — The intramuscular dose (0.5 mL contains 15 micrograms antigen from each strain and the intradermal doses (2 x 0.1 mL)contain 6 micrograms antigen from each strain.
  Other Names: Influenza vaccine

SUMMARY:
The influenza virus, commonly called the flu, is a common source of infection in lung transplant patients and can often lead to pneumonia and possibly rejection. The annual influenza vaccine is the most important strategy used to prevent infection but it is not effective in all lung transplant patients. It has been thought that the response to the vaccine may be improved if it is given into the skin (intradermal) rather than the muscle (intramuscular). We hypothesize that a significantly greater proportion of patients will respond to vaccination using the intradermal influenza vaccine compared to the intramuscular vaccine.

DETAILED DESCRIPTION:
The annual influenza vaccine is suggested for immunocompromised patients. However, the immunogenic response to this vaccine is suboptimal and ranges from 15-70%. In lung transplant recipients, responses to the influenza vaccine are poorest of all organ transplant groups. For example, a study with 43 stable lung transplant recipients showed that protective antibody developed in 19%, 30%, and 40% for the three antigens in the vaccine (only 8.6% of subjects developed protective antibody levels against all three). Similarly, 43% responded after a single dose of vaccine was given to 68 lung transplant recipients; response was significantly lower in those on mycophenolate mofetil (MMF). We have recently published a study in 60 lung transplant recipients where the standard influenza vaccine was immunogenic to at least one vaccine antigen in approximately 60% of the patients.

The study we propose is a prospective randomized control trial designed to assess the immunogenicity of the influenza vaccine given intradermally compared to the standard intramuscular vaccine in lung transplant recipients. Lung transplant recipients are unique in that their vaccine responses are the lowest of all organ groups and they stand to benefit most from an alternate vaccine strategy.

CLINICAL SIGNIFICANCE OF THE STUDY Lung transplant recipients appear to have one of the poorest humoral responses to influenza vaccination of all the organ transplant groups. However, influenza remains an important cause of morbidity in this population in whom protection is imperative. The current vaccine is suboptimal and newer strategies need to be studied to increase response rates. This subject area is of critical importance to study and especially in light of the threat of pandemic influenza.

OBJECTIVE AND HYPOTHESIS

* To test the specific humoral and cellular response after the intradermal influenza vaccine.
* To test the safety of the intradermal influenza vaccine in the lung transplant population.
* We hypothesize that a significantly greater proportion of patients will respond to vaccination using the intradermal influenza vaccine compared to the intramuscular vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Greater than 3 months post-transplant
* Outpatient status

Exclusion Criteria:

* Has already received influenza vaccination for 2008-2009 season
* Egg allergy
* Previous life-threatening reaction to influenza vaccine (i.e. Guillain Barre Syndrome)
* On anticoagulants such as warfarin that precludes intramuscular injection
* Ongoing therapy for rejection
* Febrile illness in the past two weeks
* Unable to provide informed consent
* Unable to comply with study protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2008-10; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Seroconversion rate: serological response with a four-fold or greater increase in HI antibody titers Seroprotection rate: HIA titers of >/= 1:40 | 4 weeks

SECONDARY OUTCOMES:
Local and systemic adverse events to vaccination | 24 hours, 48 hours and 7 days after each vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Deepali Kumar, Msc, FRCPC, Principal Investigator — University of Alberta
Locations (2):
- University of Alberta Hospital, Edmonton, Alberta, Canada
- University Hospital of Lausanne, Lausanne, Switzerland

REFERENCES:
- [Result] Manuel O, Humar A, Chen MH, Chernenko S, Singer LG, Cobos I, Kumar D. Immunogenicity and safety of an intradermal boosting strategy for vaccination against influenza in lung transplant recipients. Am J Transplant. 2007 Nov;7(11):2567-72. doi: 10.1111/j.1600-6143.2007.01982.x. Epub 2007 Oct 1. PMID 17908277
- See also: The Centers for Disease Control and Prevention (CDC) and the Canadian National Advisory Committee on Immunization (NACI) currently recommends this vaccine for children > 6 months, healthy adults, the elderly and all immunocompromised patients — http://www.cdc.gov